CLINICAL TRIAL: NCT03377218
Title: Safety and Efficacy of Iodine Supplementation During Pregnancy With and Without Selenium Co-administration: Randomized Controlled Trial
Brief Title: Potential Preventive Effect of Selenium on Iodine-induced Thyroid Autoimmunity During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riga Stradins University (Other)
Collaborators: Latvian Biomedical Research and Study Centre (Other Government); Riga Maternity hospital (Unknown); Latvian Institute of Organic Synthesis (Other)
Responsible Party: Principal Investigator, Ilze Konrade, associate professor, Riga Stradins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RigaStradinsU_Iodine3
Record Dates: First submitted 2017-11-18; First posted 2017-12-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Pregnancy; Thyroid Autoimmune Disease; Iodine Deficiency; Selenium Deficiency
MeSH Terms: interventions — Iodine; Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Without additional iodine supplementation.
- Iodine (Experimental): Receiving iodine.
  Interventions: Dietary Supplement: Iodine
- Iodine + Selenium (Experimental): Receiving iodine and selenium.
  Interventions: Dietary Supplement: Iodine + Selenium

INTERVENTIONS:
Dietary Supplement: Iodine — Receiving 150 μg iodine (as potassium iodide) daily
  Arms: Iodine
Dietary Supplement: Iodine + Selenium — Receiving a combination of 150 μg iodine (as potassium iodide) and 100 μg selenium daily
  Arms: Iodine + Selenium

SUMMARY:
In 1994, the WHO and UNICEF Joint Committee on Health Policy recommended Universal Salt Iodization as a safe, cost-effective and sustainable strategy to ensure sufficient intake of iodine by all individuals. However, it is still absent in Latvia.

A recent countrywide study in 2013 shows iodine deficiency among pregnant women in Latvia: 81 % of pregnant women had UIC levels below the WHO recommended range of 150-250 mcg/g Cr.

Because mild to moderate iodine deficiency during pregnancy can adversely affect fetal brain development, WHO-UNICEF and ICCIDD advise an increase in the recommended daily dosage of iodine to 250 mcg/day for pregnant women and breastfeeding women and 150 mcg/day for women in the preconception period.

Data from a survey of the Latvian population indicate that approximately 100 mcg of iodine per day is consumed through foods and iodized salt. To meet the increased iodine requirement in pregnancy, pregnant women should take a supplement containing 150 mcg of iodine daily from the earliest time possible.

A sudden increase in iodine intake in an iodine-deficient population may increase thyroid autoimmunity. It is evident that thyroid disease has multiple adverse effects during pregnancy and in the developing fetus especially in women with elevated serum anti-thyroid antibody titers.

Studies have considered supplementing with selenium to reduce the risk of auto-immune thyroiditis/post-partum autoimmune thyroid disease. Of the 11 trials of selenium supplementation in patients with autoimmune thyroiditis, 7 have shown benefit with treatment for 6 months or longer.

Aim of study is to approve that 150 mcg of iodine daily improves iodine status in pregnant women and iodine 150 mcg in combination with selenium 100 mcg daily reduce risk of thyroid autoimmunity.

Hypothesis of study is that 150 mcg iodine daily during pregnancy improves iodine status. Iodine in combination with selenium is less associated with thyroid autoimmunity.

Study design: Pregnant women are randomized for either 150 mcg iodine intake daily or 150 mcg iodine combined with 100 mcg selenium daily. Interventional group is compared with controls without particular iodine supplementation.

Participants are asked to complete a questionnaire on dietary habits concerning iodine. Thyroid function (thyroid-stimulating hormone, free thyroxine) and thyroperoxidase antibodies (TPO-Ab) and urinary iodine are measured during first, second and third trimester of pregnancy and week 8 after delivery in both, intervention and control group.

DETAILED DESCRIPTION:
In 1994, the WHO and UNICEF Joint Committee on Health Policy recommended Universal Salt Iodization as a safe, cost-effective and sustainable strategy to ensure sufficient intake of iodine by all individuals. However, universal salt iodization is still absent in Latvia.

A recent countrywide study in 2013 shows iodine deficiency among pregnant women in Latvia. The median Cr-standardized UIC was 80.8 (interquartile range (IQR) 46.1-130.6) mcg/g Cr or 69.4 (IQR 53.9-92.6) mcg/L during pregnancy, and 81 % of pregnant women had UIC levels below the WHO recommended range of 150-250 mcg/g Cr.

Because mild to moderate iodine deficiency during pregnancy can adversely affect fetal brain development, WHO-UNICEF and ICCIDD advise an increase in the recommended daily dosage of iodine to 250 mcg/day for pregnant women and breastfeeding women and 150 mcg/day for women in the preconception period.

Data from a survey of the Latvian population indicate that approximately 100 mcg of iodine per day is consumed through foods and iodized salt. To meet the increased iodine requirement in pregnancy, pregnant women should take a supplement containing 150 mcg of iodine daily from the earliest time possible.

A sudden increase in iodine intake in an iodine-deficient population may increase thyroid autoimmunity. Studies have connected induction of disease processes with thyroglobulin (Tg) iodination, because hypo-iodinated Tg did not activate T cells; however, increasing the Tg iodine content to even normal levels in vitro led to antigenicity of the molecule. It is evident that thyroid disease has multiple adverse effects during pregnancy and the postpartum period, and in the developing fetus especially in women with elevated serum anti-thyroid antibody titers.

Previous studies have considered supplementing with selenium to reduce the risk of auto-immune thyroiditis/post-partum autoimmune thyroid disease. Potential mechanisms may be related to the selenoenzyme, GPx3, removing excess H2O2 produced in the thyrocyte for the iodination of tyrosine to give thyroid hormones, thereby preventing thyrocyte damage. Additionally, selenoprotein S (SEPS1) is involved in the control of the inflammatory response in the endoplasmic reticulum. Of the 11 trials of selenium supplementation in patients with autoimmune thyroiditis, 7 have shown benefit with treatment for 6 months or longer.

Aim of study is to approve that 150 mcg of iodine daily improves iodine status in pregnant women and iodine 150 mcg in combination with selenium 100 mcg daily reduce risk of thyroid autoimmunity.

Hypothesis of study is that 150 mcg iodine daily during pregnancy improves iodine status. Iodine in combination with selenium is less associated with thyroid autoimmunity.

Study design: Pregnant women are randomized for either 150 mcg iodine intake daily or 150 mcg iodine combined with 100 mcg selenium daily. Interventional group is compared with controls without particular iodine supplementation.

Participants are asked to complete a questionnaire on dietary habits concerning iodine intake at the moment they are recruited for study, at third trimester of pregnancy and week 8 after delivery.

Thyroid function (thyroid-stimulating hormone (TSH), free thyroxine (fT4) and thyroperoxidase antibodies (TPO-Ab) measures are assessed during first, second and third trimester of pregnancy and week 8 after delivery in both, intervention and control group. Blood samples are sent to the E. Gulbis Laboratory (Riga, Latvia), which operates according to EN ISO 15189:2008 standard. TSH, fT4 and TPO-Ab are measured by chemiluminescence immunoassay (Siemens, Malvern, PA, USA).

Urinary iodine, using the ammonium persulfate method, is also measured in first, second, third trimester of pregnancy and postpartum week 8 in intervention and control groups.

The urinary creatinine concentration is measured using the Jaffe method with the intention that iodine concentration adjusted for creatinine concentration (iodine/Cr) could be calculated. Creatinine standardized UIC is a more reliable method of iodine excretion than random spot UIC measurement since there is a great day-to-day variability in water intake.

Statistical analysis includes pairwise comparison of 1) median (interquartile range) urinary iodine concentration, median (IQR) or mean (SD) TSH, and median (IQR) or mean (SD) fT4; 2) proportion (95%CI) of women with UIC below 150 mcg, TSH above trimester-specific norm, and positive TPO antibodies among all three study groups at specific follow-up intervals. Mann-Whitney U test or two-sided t-test is used for comparing continuous variables, whereas chi2 test (or Fisher exact test) is used to compare proportions. If significant differences observed at baseline, the change in those parameters from visit to visit is calculated and compared. Logistic regression analysis is used to compare intervention groups with control group in order to adjust for differences in baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

* healthy women before 10 weeks of gestation
* signed informed consent form

Exclusion Criteria:

* pre-existing thyroid disease
* pregnancy after assisted reproductive technologies
* known hypersensitivity reaction to iodine or selenium, or other components of dietary supplement used in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
UIC | At baseline - 9/10 weeks of gestation, second sample - 24 weeks of gestation (14 weeks from baseline), third sample - 34 weeks of gestation (24 weeks from the baseline) and fourth sample - 8 weeks postpartum- (38 weeks after the baseline sample)
  Urinary iodine concentration
Change in anti-TPO Ab | At baseline - 9/10 weeks of gestation, second sample - 24 weeks of gestation (14 weeks from baseline), third sample - 34 weeks of gestation (24 weeks from the baseline) and fourth sample - 8 weeks postpartum- (38 weeks after the baseline sample)
  Change in anti-thyroperoxidase antibodies

SECONDARY OUTCOMES:
TSH | At baseline - 9/10 weeks of gestation, second sample - 24 weeks of gestation (14 weeks from baseline), third sample - 34 weeks of gestation (24 weeks from the baseline) and fourth sample - 8 weeks postpartum- (38 weeks after the baseline sample)
  Thyroid stimulating hormone
fT4 | At baseline - 9/10 weeks of gestation, second sample - 24 weeks of gestation (14 weeks from baseline), third sample - 34 weeks of gestation (24 weeks from the baseline) and fourth sample - 8 weeks postpartum- (38 weeks after the baseline sample)
  Free thyroxine

CONTACTS AND LOCATIONS:
Overall Officials: Ilze Konrade, professor, Principal Investigator — Riga Stradins University
Locations (1):
- Riga Maternity hospital, Riga, Latvia